CLINICAL TRIAL: NCT04172909
Title: LEGO MRI: Decreasing the Need for Sedation, and Improving Patient Anxiety.
Acronym: LEGO MRI
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Expired IRB approval 12/12/2020
Sponsor: Montefiore Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2019-10682
Record Dates: First submitted 2019-11-10; First posted 2019-11-21 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2022-02

CONDITIONS: Stress; Anesthesia; Children, Only; Anxiety; MRI; Sedation
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: There will be two experimental groups including the LEGO Bricks group, and the Mock MRI tube group, as well as a retrospective age matched control group.
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Child life group with LEGO bricks (Experimental): Patients in this group will be prepped by a Certified Child Life Specialist with the use of LEGO bricks model MR
  Interventions: Other: LEGO Bricks MRI
- Control group (No Intervention): Age matched controls will be found retrospectively, and will be patients of the same age, undergoing their first non-contrast brain MRI with no Child Life intervention.
- Child life group with Mock MRI tube (Experimental): Patients in this group will be prepped by a Certified Child Life Specialist with the use of a Mock MRI tube
  Interventions: Other: Mock MRI tube

INTERVENTIONS:
Other: LEGO Bricks MRI — LEGO Bricks model MRI (A model of the MRI machine and adjacent control room made out of LEGO bricks) will be used by the child life specialist to prepare the child for MRI
  Arms: Child life group with LEGO bricks
Other: Mock MRI tube — Mock MRI tube will be used by the child life specialist to prepare the child for MRI
  Arms: Child life group with Mock MRI tube

SUMMARY:
The objective of the LEGO®Bricks MRI project is to study a new play-based tool for use in children preparing to undergo MRI and evaluate its ability to reduce the need for anesthesia.

A randomized study design will be employed in the experimental "Child Life" (CL) group, in regard to which Child Life intervention patients will have. Age matched controls will be found retrospectively, and will be patients of the same age, undergoing their first non-contrast brain MRI with no Child Life intervention.

Patients in the CL group will be prepped by a Certified Child Life Specialist with the use of one of the following 2 tools, to be randomly selected:

1. LEGO Bricks model MRI (A model of the MRI machine and adjacent control room made out of LEGO bricks)
2. Mock MRI tube (A six foot long pop-out play tunnel for children, with a diameter of around 17 inches to simulate the MRI magnet bore)

DETAILED DESCRIPTION:
Diagnostic imaging is frequently utilized in modern medical practice, and various imaging modalities are routinely utilized in the care of pediatric patients. Magnetic resonance imaging (MRI) is an advanced imaging modality that is utilized to evaluate many conditions in pediatric patients. MRI is frequently favored over other imaging modalities in pediatrics since it allows for high-quality cross sectional imaging without the use of potentially harmful ionizing radiation, to which children are more sensitive than adults. However, MRI quality is highly dependent on patients' ability to hold still and follow instructions, which is often challenging in pediatric patients. Young and uncooperative children often require anesthesia to successfully complete MRI. Anesthesia can often be avoided with the assistance of Certified Child Life Specialists, who use techniques to reduce patient anxiety and improve children's ability to follow instructions during MRI. For example, children may visit the MRI unit or a simulator prior to the examination to contextualize the procedure1-3. Preparation, in the form of play, has been proven to reduce anxiety in children prior to scans and invasive medical procedures. Children who are prepared for medical procedures experience less fear and anxiety and will have better long term adjustment to medical challenges (Koller, 2008).

ELIGIBILITY:
Inclusion Criteria:

* Between 4 and 10 years of age
* Undergoing first MRI
* MRI brain without contrast

Exclusion Criteria:

* Diagnosed serious illness/mental disability
* Have undergone prior MRI

Ages: 4 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2020-02-24 (Actual); Primary Completion 2022-02-01 (Estimated); Study Completion 2022-02-01 (Estimated)

PRIMARY OUTCOMES:
Number of participants who need anesthesia - Comparing CL groups ((1) LEGO Bricks model MRI and (2) mock MRI tube groups) and Control group | Up to 90 minutes (duration of MRI exam)
  Monitor whether or not the child needs anesthesia to successfully complete MRI exam

SECONDARY OUTCOMES:
Change in Anxiety Scores -Comparing CL groups (1) LEGO Bricks model MRI and (2) mock MRI tube -- Control group will not have Anxiety Scores available, and will not be assessed on this secondary outcome measure. | At time of enrollment (Baseline) and at the end of MRI exam, which typically ranges from 15-90 minutes
  Anxiety score will be measured by response to a series of questions using an anxiety self rating scale where for each questions particpants need to decide if Not at all applies (mark 1) Somewhat (mark 2) Moderately (mark 3) Very much (mark 4).
Change in quality of MRI image- Comparing CL groups ((1) LEGO Bricks model MRI and (2) mock MRI tube groups) and Control group using image quality and motion artifact grading scale | 1-2 weeks (average time to get MRI results)
  This will be assessed by blinded attending radiologist/ resident radiologist. The above mentioned grading scale scores motion artifact and image quality on a 1 to 4 and 0 to 3 scales as follows:
  Image quality:
  1 (excellent images, with very high confidence in diagnostic content), 2 (good images, with confidence in diagnostic content), 3 (fair images, with reservations about diagnostic content), 4 (poor nondiagnostic image),
  Motion artifact:
  0 (no motion artifact)
  1. (minimal motion artifact not interfering with diagnostic content)
  2. (moderate motion artifact degrading diagnostic content)
  3. (severe motion artifact resulting in non diagnostic image)
Change in duration of MRI exam-Comparing time stamp (ending time of exam minus beginning time of exam) of MRI in CL groups ((1) LEGO Bricks model MRI and (2) mock MRI tube groups) and Control group | At the end of MRI exam, which typically ranges from 15-90 minutes
  Total length of time from beginning to end of MRI scan will be recorded and compared between groups, by subtracting the start time of the exam from the end time of the exam.

CONTACTS AND LOCATIONS:
Overall Officials: Mark Liszewski, MD, Principal Investigator — Montefiore Medical Center
Locations (1):
- Montefiore Medical Center, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Saleh RS, Patel S, Lee MH, Boechat MI, Ratib O, Saraiva CR, Finn JP. Contrast-enhanced MR angiography of the chest and abdomen with use of controlled apnea in children. Radiology. 2007 Jun;243(3):837-46. doi: 10.1148/radiol.2433060155. PMID 17517937